CLINICAL TRIAL: NCT00112463
Title: A Phase II Study of Single Agent Depsipeptide (FK228) in Metastatic or Unresectable Soft Tissue Sarcomas
Brief Title: Depsipeptide (Romidepsin) in Treating Patients With Metastatic or Unresectable Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01037; NCI-2012-01037 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 71103 (Other: Wake Forest University Health Sciences); 6319 (Registry Identifier: CTEP); U10CA081851 (NIH); P30CA012197 (NIH); NCT01645683 (obsolete NCT alias)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Adult Alveolar Soft-part Sarcoma; Adult Angiosarcoma; Adult Epithelioid Sarcoma; Adult Extraskeletal Chondrosarcoma; Adult Extraskeletal Osteosarcoma; Adult Fibrosarcoma; Adult Leiomyosarcoma; Adult Liposarcoma; Adult Malignant Fibrous Histiocytoma; Adult Malignant Hemangiopericytoma; Adult Malignant Mesenchymoma; Adult Neurofibrosarcoma; Adult Rhabdomyosarcoma; Adult Synovial Sarcoma; Gastrointestinal Stromal Tumor; Metastatic Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Adult Soft Tissue Sarcoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part; Hemangiosarcoma; Sarcoma; Chondrosarcoma, Extraskeletal Myxoid; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Malignant mesenchymal tumor; Neurofibrosarcoma; Rhabdomyosarcoma; Sarcoma, Synovial; Gastrointestinal Stromal Tumors; Neuroectodermal Tumors, Primitive, Peripheral | interventions — romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (single-agent depsipeptide) (Experimental): Patients receive depsipeptide (romidepsin) intravenously (IV) over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 6 additional courses beyond documentation of CR.
  Interventions: Drug: romidepsin

INTERVENTIONS:
Drug: romidepsin — DEP is administered at a dose of 13 mg/m2 as a 4-hour intravenous infusion in the outpatient setting.
  Other Names: FK228; FR901228; Istodax

SUMMARY:
This phase II trial studies how well depsipeptide (romidepsin) works in treating patients with metastatic or unresectable soft tissue sarcoma. Drugs used in chemotherapy, such as depsipeptide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the response rates of metastatic or unresectable soft tissue sarcomas to single-agent depsipeptide.

II. To estimate the time to progression of metastatic or unresectable soft tissue sarcomas to single-agent depsipeptide.

III. To evaluate the scope and extent of acute toxicities associated with single-agent depsipeptide when given to patients with soft tissue sarcomas.

OUTLINE: This is a multicenter study.

Patients receive depsipeptide (romidepsin) intravenously (IV) over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 6 additional courses beyond documentation of CR.

After completion of study treatment, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed soft tissue sarcoma (STS), including, but not limited to, the following histologies:

  * Gastrointestinal stromal tumors (GIST)

    * Refractory to imatinib mesylate
  * Desmoplastic small round cell tumors
  * Clear cell sarcoma
  * Extraskeletal osteosarcoma*
  * Extraskeletal Ewing's sarcoma*
  * Extraskeletal (myxoid) chondrosarcoma*
* Secondary STS (e.g., radiation-induced STS or neurofibrosarcoma due to neurofibromatosis) allowed
* Metastatic or unresectable disease
* No standard curative therapy exists
* Patients with GIST must have received and progressed on imatinib mesylate
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No known brain metastases
* Performance status - Eastern Cooperative Oncology Group (ECOG) 0-2
* Performance status - Karnofsky 50-100%
* More than 3 months
* White blood cells (WBC) â¥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) â¤ 2.5 times upper limit of normal (ULN)
* Bilirubin normal
* Creatinine < 1.5 times ULN
* Creatinine clearance ≥ 60 mL/min
* QTc ≤ 480 msec

Exclusion Criteria:

* No cardiac abnormalities (e.g., congenital long QT syndrome)
* No myocardial infarction within the past year
* No history of coronary artery disease (e.g., angina Canadian Class II-IV or positive stress imaging study)
* No cardiac ischemia (ST depression >2 mm) by electrocardiogram (ECG)
* No New York Heart Association Class II-IV congestive heart failure
* Ejection fraction > 50% by multi gated acquisition scan (MUGA) scan or echocardiogram
* No history of sustained ventricular tachycardia, ventricular fibrillation, Torsades de Pointes, or cardiac arrest unless controlled by an automatic implantable cardioverter defibrillator
* No hypertrophic or restrictive cardiomyopathy from prior treatment or other causes
* No significant left ventricular hypertrophy
* No uncontrolled hypertension (i.e., blood pressure ≥ 160/95 mm Hg)
* No cardiac arrhythmia requiring anti-arrhythmic medication

  * Beta blocker or calcium channel blocker allowed
  * Patients on digitalis that cannot be discontinued not allowed
* No Mobitz II second degree block without a pacemaker (first degree or Mobitz I second degree block, bradyarrhythmias, or sick sinus syndrome require Holter monitoring and evaluation by cardiology)
* No uncontrolled dysrhythmia
* No poorly controlled angina
* No other cardiac disease
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to FR901228
* No ongoing or active infection
* No iatrogenic immune deficiency or immune deficiency secondary to an underlying disorder
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Potassium ≥ 4.0 mmol/L
* Magnesium ≥ 2.0 mg/dL
* No other uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No concurrent anticancer biologic agents
* No more than 1 prior chemotherapy regimen for sarcoma

  * Adjuvant chemotherapy preceding disease relapse is considered 1 prior chemotherapy regimen
  * Patients with GIST may have received up to 3 prior chemotherapy regimens comprising imatinib mesylate and/or sunitinib malate provided no other chemotherapy agents were used
* No prior FR901228 (depsipeptide)
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No prior cumulative doxorubicin dose > 500 mg/m^2
* No other concurrent anticancer chemotherapy
* At least 4 weeks since prior radiotherapy
* No concurrent anticancer radiotherapy
* At least 4 weeks since prior surgery
* No prior organ transplantation
* Recovered from all prior therapy
* No concurrent medications that cause QTc prolongation
* No concurrent combination highly active anti-retroviral therapy for HIV-positive patients
* No other concurrent drugs known to have histone deacetylase inhibitor activity (e.g., sodium valproate)
* No other concurrent investigational agents
* No other concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-01-07 (Actual); Primary Completion 2008-10-23 (Actual); Study Completion 2008-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Savage, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Single-agent Depsipeptide)
Started | 40
Completed | 1
Not Completed | 39
Not completed — Physician Decision | 1
Not completed — Progression | 30
Not completed — Second Primary | 1
Not completed — Toxicity | 3
Not completed — Withdrawal by Subject | 2
Not completed — Never started treatment | 2

BASELINE CHARACTERISTICS:
Population: All registered participants
Arm/Group | Treatment (Single-agent Depsipeptide)
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 16
Age, Continuous [Median (Full Range); unit: years] | 59 [19 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 32
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response (Complete and Partial)
Description: Objective tumor response was evaluated using the criteria proposed by the Response Evaluation Criteria In Solid Tumors (RECIST) Committee (JNCI 92(3):205-216,2000). Changes in only the largest diameter (unidimensional measurement) of the target lesions are used. A sum of the longest diameter (LD) for all target lesions was calculated and reported as the baseline sum LD. The baseline sum LD was used as reference by which to characterize the objective tumor response. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum LD; Overall Response (OR) = CR + PR
Time Frame: While on treatment - max of 16 months
Population: Participants who were evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Single-agent Depsipeptide)
Number analyzed (Participants) | 35
Participants | 2

2. Primary Outcome: Time to Progression
Description: Progressive disease is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameters (LD) of target lesions, taking as reference the smallest sum LD recorded since treatment started, or a measurable increase in a non-target lesion, or the appearance of new lesions. Time to progression is the number of months from first treatment until the date of progression.
Time Frame: Until disease progression - max of 48 months
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Single-agent Depsipeptide)
Number analyzed (Participants) | 38
months | 1.9 [1.7 to 2.5]

3. Primary Outcome: Toxicity as Assessed Using the Expanded Common Toxicity Criteria Version 3
Description: The outcome reported here is the number (%) of participants who experienced grade 3 or greater toxicity while on study.
  A summary of the individual toxicities can be found in the AE/SAE results.
Time Frame: During treatment (max of 16 months) and for 1 month following treatment
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Single-agent Depsipeptide)
Number analyzed (Participants) | 38
Participants | 13

4. Secondary Outcome: Survival
Description: Months from first treatment until death or the last date of contact
Time Frame: Max of 98 months
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Single-agent Depsipeptide)
Number analyzed (Participants) | 38
months | 12.2 [7.6 to 19.3]

ADVERSE EVENTS:
Time Frame: During treatment (max of 16 months) and for 1 month following treatment
Description: Toxicities were evaluated weekly while the participant was on treatment
Arm/Group | Treatment (Single-agent Depsipeptide)
Serious Adverse Events (participants affected / at risk) | 13/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Single-agent Depsipeptide) (N=38)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Cardiac Arrhythmia - Other (Cardiac disorders) | 3 (4)
Cardiac Dysrhythmia (Cardiac disorders) | 1 (1)
Cardiac General - Other (Cardiac disorders) | 2 (2)
Coagulation - Other (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
GI - Other (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 2 (3)
Infection - Other (Infections and infestations) | 1 (1)
Malise/Fatigue (Metabolism and nutrition disorders) | 1 (1)
Metabolic - Other (Metabolism and nutrition disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 3 (5)
Pain - Other (Nervous system disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 4 (5)
Weight Loss (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Single-agent Depsipeptide) (N=38)
AGC/ANC (Immune system disorders) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 9 (55)
Cardiac Arrhythmia (Cardiac disorders) | 5 (9)
Caridac General - Other (Cardiac disorders) | 4 (4)
Coagulation - Other (Blood and lymphatic system disorders) | 3 (5)
Constipation (Gastrointestinal disorders) | 19 (82)
Constitutional Symptioms - Other (Gastrointestinal disorders) | 13 (51)
Creatinine (Renal and urinary disorders) | 3 (3)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 6 (11)
Diarrhea (Gastrointestinal disorders) | 8 (9)
Dizziness (Nervous system disorders) | 3 (16)
Dyspepsia/Heartburn (Gastrointestinal disorders) | 4 (20)
Dyspnea/SOB (Respiratory, thoracic and mediastinal disorders) | 14 (26)
Fever in the absence of neutropenia (Infections and infestations) | 3 (4)
GI - Other (Gastrointestinal disorders) | 25 (65)
Hemoglobin (Blood and lymphatic system disorders) | 11 (84)
Hot flashes/flushes (Endocrine disorders) | 3 (19)
Hyperglycemia (Endocrine disorders) | 5 (14)
Infection - Other (Infections and infestations) | 6 (10)
Malise/Fatigue (Metabolism and nutrition disorders) | 32 (198)
Metabolic - Other (Metabolism and nutrition disorders) | 9 (21)
Mucositis/stomatitis (Infections and infestations) | 4 (6)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (8)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 11 (23)
Nausea (Gastrointestinal disorders) | 26 (150)
Neurologic - Other (Nervous system disorders) | 14 (59)
Pain - Other (Nervous system disorders) | 22 (123)
Pain: Abdomen NOS (Nervous system disorders) | 3 (8)
Pain: Back (Nervous system disorders) | 4 (5)
Pain: Extremity-limb (Nervous system disorders) | 4 (15)
Pain: Head/Headache (Nervous system disorders) | 4 (5)
Pain: NOS (Nervous system disorders) | 7 (22)
Pulmonary Other (Respiratory, thoracic and mediastinal disorders) | 7 (18)
Renal/Genitourinary - Other (Renal and urinary disorders) | 5 (7)
Taste Alteration (Nervous system disorders) | 7 (49)
Vomiting (Gastrointestinal disorders) | 15 (42)
WBC (Infections and infestations) | 4 (11)
Weight Gain (Metabolism and nutrition disorders) | 3 (3)
Weight Loss (Metabolism and nutrition disorders) | 11 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less